CLINICAL TRIAL: NCT02513862
Title: Prospective Randomized Trial of Autologous Platelet Rich Plasma in Reducing Allogeneic Transfusions During Aortic Surgery Under Deep Hypothermic Circulatory Arrest
Brief Title: Prospective Trial of Autologous Platelet Rich Plasma in Aortic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hongwen Ji (Other)
Responsible Party: Sponsor-Investigator, Hongwen Ji, professor of medicine, Chinese Academy of Medical Sciences, Fuwai Hospital
Organization: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2014-zx011
Record Dates: First submitted 2015-06-23; First posted 2015-08-03 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2016-11

CONDITIONS: C.Surgical Procedure; Cardiac
Keywords: autologous platelet rich plasma; deep hypothermic circulatory arrest; transfusion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- APRP group (Experimental): APRP group is performed autologous platelet-rich plasma harvest technique before administration of heparin to the patient,the red blood cell(RBC) component is retransfused to the patient when the RBC transfusion protocol is reached,and the autologous platelet-rich plasma is transfused to the patient immediately after heparin is neutralized with protamine.
  Interventions: Device: Autologous Platelet-Rich Plasma Harvest Technique
- control group (No Intervention): APRP group receive no autologous platelet-rich plasma harvest technique.

INTERVENTIONS:
Device: Autologous Platelet-Rich Plasma Harvest Technique — 15 to 20 mL/kg of whole blood is collected before the administration of heparin from a large-bore central venous access,and is separated into red blood cells component and autologous platelet-rich plasma component by an autologous transfusion system(Sorin Group Electa Essential; Sorin Group Italia, Milan, Italy).
  Other Names: neutralizing heparin with protamine
  Arms: APRP group

SUMMARY:
The purpose of this study is to determine whether autologous platelet rich plasma (APRP)is effective in reducing allogeneic blood transfusions during aortic surgery using deep hypothermic circulatory arrest.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective or emergency aortic surgery using deep hypothermic circulatory arrest、
* preoperative platelet counts>150000000000/L、
* preoperative hematocrit>33%、
* without recent anticoagulants less than 5 days

Exclusion Criteria:

* preoperative coagulation disorder
* severe renal and liver dysfunction
* preoperative hemodynamic instability

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-05; Primary Completion 2016-06 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
total perioperative allogenic transfusions of platelet and fresh frozen plasma | on the 7th day postoperatively

SECONDARY OUTCOMES:
postoperative blood loss | on the 7th day postoperatively
rate of reexploration for bleeding | on the 7th day postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Hongwen Ji, MD, Study Chair — Cardiovascular Institute and Fuwai Hospital, CAMS&PUMC; Yongyuan Wang, Principal Investigator — Cardiovascular Institute and Fuwai Hospital, CAMS&PUMC
Locations (1):
- Cardiovascular Institute and Fuwai Hospital, CAMS&PUMC, Beijing, Beijing Municipality, China